CLINICAL TRIAL: NCT02281045
Title: CITrate and Evodial for Effective Dialysis (CITED) Study
Acronym: CITED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S55895
Record Dates: First submitted 2014-10-22; First posted 2014-11-03 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVODIAL dialyzer and Selectbag citrate (Experimental): Intervention for anticoagulation during dialysis: Combination of Heparin-coated AN69ST membrane (EVODIAL, Gambro-Hospal, Meyzieu, France) and citrate-containing dialysate (Selectbag citrate, Gambro, Lund, Sweden).
  Interventions: Device: EVODIAL dialyzer and Selectbag citrate
- Regional citrate anticoagulation (Active Comparator): Regional citrate anticoagulation, using a hypertonic sterile solution of trisodium citrate dihydrate (1.035 Mol/L, Baxter, Lessines, Belgium), infused into the afferent blood line. Citrate will be infused at a rate of 62.1 mM/h (60 mL/h). The anticoagulant effect of citrate will be neutralized using calcium containing dialysate (Ca 1.50 mmol/L). Dialysate sodium content will be set at 135 mEQ/L, and bicarbonate will be reduced to 25 mEq/L.
  Interventions: Device: Regional citrate anticoagulation

INTERVENTIONS:
Device: EVODIAL dialyzer and Selectbag citrate — Evodial is a trademark of Hospal-Gambro.
  Arms: EVODIAL dialyzer and Selectbag citrate
Device: Regional citrate anticoagulation — Regional citrate anticoagulation is performed according to local practice, using a calcium-containing dialysate
  Arms: Regional citrate anticoagulation

SUMMARY:
It is not known whether the combination of a heparin-grafted membrane plus citrate-containing dialysate is a valid alternative to regional citrate anticoagulation. This is a cross-over non-inferiority trial comparing these two anticoagulation strategies

DETAILED DESCRIPTION:
Anticoagulation is one of the supporting pillars of chronic hemodialysis (HD) (1). The optimal anticoagulant regimen provides full anticoagulation of the extracorporeal circuit with minimal systemic effects and comes at an affordable cost. Unfractionated heparin (UFH) has been the standard of care for many years. In several countries, UFH has gradually been replaced by low molecular weight heparins (LMWH). LMWH are easy to use as they can be administered as a bolus injection and reduce membrane fibrin and platelet deposition (2,1). Both UFH or LMWH provide adequate anticoagulation of the extracorporeal circuit, at the price of systemic anticoagulation. Apart from bleeding, the administration of unfractionated heparins has also been associated with dyslipidemia, hypoaldosteronism and hyperkalemia, thrombopenia, osteoporosis, pruritus, and hypersensitivity reactions.

Several alternative anticoagulation regimens have been proposed including heparin coating of the dialyzer membrane and regional citrate anticoagulation. Regional citrate anticoagulation is performed by infusing citrate into the arterial line of the dialysis tubing to reduce ionized calcium concentrations to very low levels (4,1). Ionized calcium concentrations are restored by calcium supplementation prior to reinfusion of the blood into the patient. Most often, calcium repletion is by calcium infusion into the venous line. Alternatively, a conventional calcium containing dialysate will restore calcium concentrations and, although the anticoagulant effect is blunted in the venous line, gives acceptable results (5). A previous study suggested that regional citrate anticoagulation is superior to heparin-coated polyacrylonitrile dialyzers (AN69ST; Nephral 300ST, Gambro) and resulted in in significantly greater instantaneous urea nitrogen clearances (3).

While generally safe and adequate, regional citrate anticoagulation requires additional actions during preparatory phase (preparation of citrate and calcium infusion pumps) as well as during the treatment (measurement of ionized calcium). These additional actions result in additional costs.

Recently, acetate-free citrate-containing dialysate concentrates were introduced into clinical practice. Besides the advantages of acetate-free dialysate, this provides a modest local anticoagulant effect inside the dialyzer. Citrate-containing dialysate allowed to reduce heparin dose while maintaining extracorporeal circuit patency and dialyzer clearances (6).

The investigators questioned whether combination of citrate-containing dialysate and heparin-coated dialyzer membranes is equally effective as conventional regional citrate anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years,
* hemodynamic stability,
* hemoglobin 9 - 12 g/dl.

Exclusion Criteria:

* Any hemostatic disorder favoring either bleeding or clotting,
* anti-vitamin K treatment,
* risk of bleeding according to the criteria of Swartz (12).

Treatment with aspirin, dipyridamole or any drugs likely to interfere with platelet aggregation will be registered carefully, but will not be an exclusion criterion.

All vascular access types (AV-fistula, AV graft, catheter) are allowed. However, only patients with double route vascular access ('bipuncture') will be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Patency of hemodialysis circuit | 20 weeks
  Completion of 4h dialysis session without circuit clotting that requires early treatment interruption

SECONDARY OUTCOMES:
Clotting of dialyser after the rinse | 20 weeks
  scored semi-quantitatively on a visual scale (0: no clotting; 1: mild clotting; 2: severe clotting, 4: completely clotted).

CONTACTS AND LOCATIONS:
Overall Officials: Björn Meijers, MD, PhD, Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593